CLINICAL TRIAL: NCT05990127
Title: A Randomized, Double-blind, Phase III Trial to Compare the Efficacy and Safety of AK104 Combined With Chemotherapy to Tislelizumab Combined With Chemotherapy as First-line Treatment in PD-L1 TPS < 1% Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Study of AK104/Tislelizumab With Chemotherapy as First-line Treatment in PD-L1 TPS < 1% Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-307
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 arm (Experimental)
  Interventions: Drug: AK104; Drug: carboplatin; Drug: Pemetrexed; Drug: Paclitaxel
- Tislelizumab arm (Active Comparator)
  Interventions: Drug: Tislelizumab; Drug: carboplatin; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: AK104 — AK104 IV, q3w
  Arms: AK104 arm
Drug: Tislelizumab — Tislelizumab IV, q3w
  Arms: Tislelizumab arm
Drug: carboplatin — carboplatin IV, q3w
Drug: Pemetrexed — Pemetrexed IV, q3w (for Nonsquamous NSCLC)
Drug: Paclitaxel — Paclitaxel IV, q3w (for squamous NSCLC)

SUMMARY:
This is a randomized, double-blind, phase III clinical study to compare the efficacy and safety of AK104 combined chemotherapy versus Tislelizumab combined chemotherapy in first-line treatment of Locally advanced or metastatic NSCLC with PD-L1 TPS < 1%.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study with full informed consent and signed written informed consent form.
2. Aged ≥18 years when the subject signed the informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy ≥ 3 months.
5. Histologically or cytologically confirmed locally advanced (Stage IIIB/IIIC) that not amenable to complete surgical resection and not amenable to radical concurrent/sequential chemoradiation or metastatic (Stage IV) NSCLC (American Joint Committee on Cancer [AJCC] 8th edition).
6. No prior systemic therapy for advanced or metastatic NSCLC was received.
7. PD-L1 TPS < 1%.
8. No EGFR sensitive mutations or ALK gene translocation alterations.

Exclusion Criteria:

1. Histologically confirmed small cell lung cancer (SCLC).
2. NSCLC with driver gene mutations for approved targeted drug indications.
3. Active central nervous system (CNS) metastases were present.
4. Pulmonary radiation therapy > 30 Gy within 6 months prior to first dose.
5. Active malignant tumors within the past 5 years, except for tumors in this study and scured local tumors.
6. Pregnant or lactating women.
7. Clinically significant cardiovascular or cerebrovascular disease.
8. Subjects with a known history of severe hypersensitivity to other monoclonal antibodies. A known history of allergy or hypersensitivity to all investigational drugs or any of their components.
9. Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment, or autoimmune diseases that may relapse or require scheduled treatment as judged by the Investigator.
10. Known active pulmonary tuberculosis.
11. Patients with active hepatitis B or active hepatitis C.
12. Known medical history of immunodeficiency or positive HIV test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Estimated)
Dates: Start 2023-11-14 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2026-11-28 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | Through Database Cutoff Date (Up to approximately 39 months)
  OS is defined as the time from randomization to death due to any cause.
Progression-Free Survival(PFS) by investigator(INV) | Through Database Cutoff Date (Up to approximately 39 months)
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1

SECONDARY OUTCOMES:
Progression-Free Survival(PFS) by Blind independent center review(BIRC) | Through Database Cutoff Date (Up to approximately 39 months)
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1
Objective response rate (ORR) was assessed by INV | Through Database Cutoff Date (Up to approximately 39 months)
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1
Disease control rate (DCR) was assessed by INV | Through Database Cutoff Date (Up to approximately 39 months)
  Disease control rate (DCR) was assessed based on RECIST V1.1 criteria
Time to response (TTR) was assessed by INV | Through Database Cutoff Date (Up to approximately 39 months)
  The time from the first administration to the date of documented CR or PR
Duration of response (DOR) was assessed by INV | Through Database Cutoff Date (Up to approximately 39 months)
  Measured from the date of partial or complete response to therapy until the disease progression per RECIST v1.1 criteria
Objective response rate (ORR) was assessed by BIRC | Through Database Cutoff Date (Up to approximately 39 months)
  ORR is the proportion of subjects with CR or PR based on RECIST v1.1
Disease control rate (DCR) was assessed BIRC | Through Database Cutoff Date (Up to approximately 39 months)
  Disease control rate (DCR) was assessed based on RECIST V1.1 criteria
Time to response (TTR) was assessed by BIRC | Through Database Cutoff Date (Up to approximately 39 months)
  The time from the first administration to the date of documented CR or PR
Duration of response (DOR) was assessed by BIRC | Through Database Cutoff Date (Up to approximately 39 months)
  Measured from the date of partial or complete response to therapy until the disease progression per RECIST v1.1 criteria
The number of subjects experiencing adverse events (AEs) | Through Database Cutoff Date (Up to approximately 39 months)
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.
Pharmacokinetic | Through Database Cutoff Date (Up to approximately 39 months)
  The endpoints for assessment of PK of AK104 include serum concentrations of AK104 at different timepoints after AK104 administration
Antidrug antibodies (ADA) of AK104 | Through Database Cutoff Date (Up to approximately 39 months)
  Proportion of subjects who develop detectable anti-drug antibodies (ADAs)
Health-related Quality of Life (HRQoL) assessment using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Through Database Cutoff Date (Up to approximately 39 months)
  EORTC QLQ-C30 measures cancer patients' physical, psychological, and social functions. Scale ranges from: 1, "Not at all"; 2, "A little"; 3, "Quite a bit"; to 4, "Very much". Higher score for the functioning scales and global health status denotes a better level of functioning, while higher scores on the symptom and single-item scales indicate a higher level of symptoms.
Health-related Quality of Life (HRQoL) assessment using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 29 module (EORTC QLQ-LC29) | Through Database Cutoff Date (Up to approximately 39 months)
  EORTC-QLQ-LC29 measures the quality of life in patients with lung cancer. Symptom scale ranges from: 1, "Not at all"; 2, "A little"; 3, "Quite a bit"; to 4, "Very much". For symptoms scales, higher scores indicated greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, M.D., Principal Investigator — Cancer hospital, Chinese academy of medical sciences and Peking union medical college; Qingming Wang, Principal Investigator — Henan Cancer Hospital
Locations (62):
- China (62):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Anhui provincial hospital, Hefei, Anhui
  - Anhui provincial cancer hospital, Hefei, Anhui
  - The first affiliated hospital of wannan medical college, Wuhu, Anhui
  - Cancer hospital, Chinese academy of medical sciences and Peking union medical college, Beijing, Beijing Municipality
  - The Fifth Medical Center of the Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian cancer hospital, Fuzhou, Fujian
  - Zhangzhou municipal hospital of fujian province, Zhangzhou, Fujian
  - Gansu provincial cancer hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated cancer hospital and institute of guangzhou medical university, Guangzhou, Guangdong
  - Nanfang hospital, Guangzhou, Guangdong
  - Cancer hospital Chinses academy of medical sciences， shenzhen center, Shenzhen, Guangdong
  - Hainan cancer hospital, Haikou, Hainan
  - Affiliated hospital of Hebei university, Baoding, Hebei
  - The second people's hospital of Hengshui, Hengshui, Hebei
  - The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshang people's hospital, Tangshan, Hebei
  - Harbin medical university cancer hospital, Harbin, Heilongjiang
  - Jiamusi Tuberculosis Prevention and Control Hospital (Jiamusi Cancer Hospital), Jiamusi, Heilongjiang
  - The first hospital of Qiqihar, Qiqihar, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang central hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The affiliated hospital of xuzhou medical university, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan medical college, Ganzhou, Jiangxi
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin Universit, Changchun, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - The First Hospital of China medical University, Shenyang, Liaoning
  - Liaoning cancer hospital, Shenyang, Liaoning
  - General hospital of ningxia medical university, Yinchuan, Ningxia
  - Qinghai university affiliated hospital, Xining, Qinghai
  - Binzhou medical university hospital, Binzhou, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang NO.2 people's Hospital, Weifang, Shandong
  - Zhongshan Hospital, Fudan university, Shanghai, Shanghai Municipality
  - Changzhi people's hospital, Changzhi, Shanxi
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Mianyang central hospital, Mianyang, Sichuan
  - The Second People's Hospital of Yibin City, Yibin, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital /the Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No